CLINICAL TRIAL: NCT07105878
Title: Epidural Electrical Stimulation for Motor and Sensory Function Reconstruction in Spinal Cord Injury
Brief Title: Epidural Electrical Stimulation in Spinal Cord Injury
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Collaborators: College of Biomedical Engineering and Instrumentation Science, Zhejiang University (Unknown)
Responsible Party: Principal Investigator, Junming Zhu, Chief Physician, Second Affiliated Hospital, School of Medicine, Zhejiang University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025-1040
Record Dates: First submitted 2025-07-30; First posted 2025-08-06 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-07

CONDITIONS: Spinal Cord Injuries (SCI)
Keywords: Epidural Electrical Stimulation; Spinal Cord Injuries; Sensor function reconstruction; Motor function reconstruction
MeSH Terms: conditions — Spinal Cord Injuries | interventions — Diffusion Tensor Imaging; Evoked Potentials, Somatosensory; Evoked Potentials, Motor

STUDY DESIGN:
Intervention Model Description: One group of patients with spinal cord injury received EES treatment and 6 months of standardized rehabilitation therapy, while the other group received only standardized rehabilitation therapy.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Epidural Electrical Stimulation (EES) + Standard Rehabilitation (Experimental): Participants receive the EES intervention combined with standard rehabilitation therapy (e.g., physical therapy, occupational therapy) for 6 months.
  Interventions: Procedure: Epidural Electrical Stimulation; Procedure: Standard Rehabilitation Therapy; Radiation: positron emission tomography-computed tomography (PET-CT); Radiation: Diffusion Tensor Imaging (DTI); Procedure: Somatosensory Evoked Potentials (SEPs); Procedure: Motor Evoked Potentials (MEPs)

INTERVENTIONS:
Procedure: Epidural Electrical Stimulation — Epidural Electrical Stimulation (EES) is a medical technology that involves delivering controlled electrical impulses to the spinal cord through electrodes implanted in the epidural space-the area between the outermost membrane of the spinal cord (dura mater) and the vertebrae. This technique aims to modulate the activity of spinal neural networks, thereby regulating neurological functions and promoting functional recovery, particularly in individuals with spinal cord injuries or certain neurological disorders.
Procedure: Standard Rehabilitation Therapy — A structured, multidisciplinary rehabilitation program designed to improve motor function, mobility, and independence in participants with paralysis. The therapy typically includes physical Therapy and occupational Therapy.
Radiation: positron emission tomography-computed tomography (PET-CT) — PET-CT is an advanced hybrid imaging modality that combines metabolic information from positron emission tomography with anatomical details from computed tomography.
Radiation: Diffusion Tensor Imaging (DTI) — DTI is an advanced MRI technique that maps white matter tracts by measuring the directionality (anisotropy) and magnitude of water molecule diffusion in neural tissues. It provides quantitative metrics of fibers.
Procedure: Somatosensory Evoked Potentials (SEPs) — SEPs are electrophysiological responses recorded from the central or peripheral nervous system following electrical stimulation of sensory nerves. They assess the functional integrity of somatosensory pathways.
Procedure: Motor Evoked Potentials (MEPs) — MEPs are electrophysiological responses elicited by transcranial magnetic stimulation or electrical stimulation of the motor cortex, recorded from peripheral muscles or the spinal cord. They evaluate the integrity of corticospinal tracts.

SUMMARY:
The goal of this clinical trial is to evaluate the safety and effectiveness of Epidural Electrical Stimulation (EES) in motor and sensory function Reconstruction in chronic spinal cord injury (SCI) patients classified as ASIA B-D. The main questions it aims to answer are:

Does EES treatment significantly improve motor and sensory function in patients with SCI compared to baseline? Is EES a safe intervention for this patient population? Researchers will compare participants' motor function, sensory function, and quality of life assessments before EES implantation, immediately after activation of the device, and at 1, 3, and 6 months post-implantation to evaluate the longitudinal effects of EES.

Participants will:

Undergo surgical implantation of an EES device in the epidural space. Have the EES device activated and receive personalized stimulation parameter adjustments during follow-up visits.

Complete regular motor and sensory function assessments using standardized protocols.

Participate in structured rehabilitation training sessions while using the EES device.

Report any adverse events and complete quality of life questionnaires at specified follow-up intervals.

ELIGIBILITY:
Inclusion Criteria:

* Spinal Cord Injury, ASIA B-D;
* Spinal cord injury level above T10;
* Diagnosed with spinal cord injury for ≥ 8 months and ≤ 36 months;
* WISCI II score < 13;
* No significant improvement in motor dysfunction after rehabitation over the past 2 months.
* An expected survival period of ≥ 12 months.
* Subjects voluntarily participate in this study, sign the informed consent form, have good compliance, cooperate with necessary postoperative rehabilitation training and tests, and assist in follow-up visits.

Exclusion Criteria:

* Subjects with other severe organic neurological diseases, mental illnesses other than anxiety/depression.
* Subjects with hemorrhagic diathesis or coagulation dysfunction (prothrombin time [PT] ≥ 18 seconds).
* Subjects with a history of alcohol or drug abuse or dependence.
* Subjects with mental retardation, cognitive dysfunction, or personality disorders.
* Subjects with a history of electroconvulsive therapy or those requiring continuous electrotherapy.
* Subjects with implanted cardiac pacemakers, cardioverters, or defibrillators. Expected survival period < 1 year.

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
WISCI II (Walking Index for Spinal Cord Injury II) | baseline, and 1, 3, 6 monthes after surgery
  The WISCI II evaluates walking ability in spinal cord injury patients. It has 21 levels (0-20), with scores based on mobility aids, assistance needed, and walking distance. A score of 0 means no walking; 20 indicates independent walking over 500 meters without aids. It tracks recovery progress and helps tailor rehabilitation plans for locomotor function.
Functional Independence Measure (FIM) | baseline, and 1, 3, 6 months after surgery
  The Functional Independence Measure (FIM) is a widely used assessment tool designed to evaluate a person's functional status and level of independence in daily living activities, particularly among individuals with disabilities.
  FIM items are scored based on the level of assistance required to complete a task, ranging from 1 to 7 points per item.
  The FIM consists of 18 items across two domains: Motor domain (13 items): Includes activities such as eating, grooming, bathing, dressing, toileting, transfers (bed/chair, toilet, tub/shower), walking, and stair climbing. Cognitive domain (5 items): Covers communication (comprehension and expression) and social cognition (memory, problem-solving, and social interaction).
  The total score ranges from 18 to 126 points:
  ≤ 35 points: Severe dependence 36-89 points: Moderate dependence 90-119 points: Mild dependence 120-126 points: Functional independence

SECONDARY OUTCOMES:
International Standards for Neurological Classification of Spinal Cord Injury (ISNCSCI) | baseline, and 1, 3, 6 monthes after surgery
  ISNCSCI is the most authoritative and widely used standard for evaluating neurological function after spinal cord injury, comprising:
  Motor Scores:
  Range:
  Upper limbs (C5-T1): 0-25 per limb (total 0-50) Lower limbs (L2-S1): 0-25 per limb (total 0-50) Total motor score: 0-100 points Higher scores indicate better motor function
  Sensory Scores:
  Light touch:
  0-2 points per dermatome (C2-S4/5) Total: 0-112 points
  Pinprick:
  0-2 points per dermatome (C2-S4/5) Total: 0-112 points Interpretation: Higher scores indicate better sensory preservation Neurological Level of Injury
  Determined by the most caudal segment with:
  ≥3/5 muscle strength (motor level) Intact sensation (sensory level) ASIA Impairment Scale (AIS)
  Grading:
  A = Complete (no motor/sensory function in S4-S5) B = Sensory incomplete C = Motor incomplete (<50% key muscles ≥3/5 below NLI) D = Motor incomplete (≥50% key muscles ≥3/5 below NLI) E = Normal
Modified Ashworth Scale | baseline, and 1, 3, 6 monthes after surgery
  The Modified Ashworth Scale (MAS) is a clinical tool used to assess muscle spasticity by grading resistance during passive movement. It scores from 0 (no tone increase) to 4 (rigid joint), with intermediate grades: 1 (slight resistance), 1+ (mild resistance through ≤50% ROM), 2 (marked resistance), and 3 (considerable resistance). Higher MAS scores (max=4) indicate worse outcomes, reflecting more severe spasticity that impairs mobility. The assessment requires standardized passive stretching at 1 joint/sec. While widely used, it shows limitations in distinguishing mild/moderate spasticity reliably.
Penn | baseline, and 1, 3, 6 months after surgery
  The Penn Scale is a specific assessment tool for measuring muscle spasticity. Scores range from 0 (no spasticity) to 4 (severe, rigid spasticity), with higher scores indicating more intense muscle stiffness and involuntary contractions.
Hamilton Depression Rating Scale (HAMD) | baseline, and 1, 3, 6 monthes after surgery
  The HAMD is a clinician-administered assessment used to measure the severity of depressive symptoms in individuals. It typically consists of 17 items, with scores based on the patient's reported feelings, behavior, and psychological state over the past week. A higher score indicates more severe depression. It is widely used to diagnose depression, evaluate treatment efficacy, and monitor symptom changes over time.
Hamilton Anxiety Rating Scale (HAMA) | baseline, and 1, 3, 6 monthes after surgery
  The HAMA is a clinician-rated scale designed to quantify the severity of anxiety symptoms. It comprises 14 items, with scores reflecting both psychic anxiety (mental agitation) and somatic anxiety (physical complaints). A higher score signifies a greater level of anxiety. It assists in diagnosing anxiety disorders, assessing their intensity, and tracking the effectiveness of therapeutic interventions.
Visual Analog Scale (VAS) | baseline, and 1, 3, 6 monthes after surgery
  The VAS Pain Score is a self-reported measure of pain intensity. It consists of a 10-cm horizontal line, anchored by "no pain" (0) on one end and "worst pain imaginable" (10) on the other. Patients mark the line to represent their current pain level, and the score is determined by measuring the distance from "no pain." It provides a simple, quick method to quantify subjective pain experiences, monitor fluctuations, and guide pain management strategies.

CONTACTS AND LOCATIONS:
Overall Officials: Junming Zhu, Chief Physician, Principal Investigator — Second Affiliated Hospital, School of Medicine, Zhejiang University
Locations (1):
- Second Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP